CLINICAL TRIAL: NCT00564382
Title: Cardiac MRI for the Diagnosis of Unstable Angina/ NSTEMI in the Emergency Room
Brief Title: CMR in the Assessment of Patient With ACS in the Emergency Room
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Oliver Strohm, adunct Research Associate Professor, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Emergency001
Record Dates: First submitted 2007-11-26; First posted 2007-11-28 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-10

CONDITIONS: Infarction; Ischemia; Magnetic Resonance Imaging
Keywords: Acute coronary syndrome; Cardiac Magnetic Resonance Imaging; Contrast agents; Gadolinium
MeSH Terms: conditions — Infarction; Ischemia; Acute Coronary Syndrome | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Patients with ACS in the emergency department and primary tests (ECG, TNT) negative for myocardial ischemia
  Interventions: Procedure: Cardiac magnetic Resonance study

INTERVENTIONS:
Procedure: Cardiac magnetic Resonance study — Routine cardiac MR study including contrast application
  Other Names: Standard of care

SUMMARY:
In this study, we investigate the role of Cardiac Magnetic Resonance Imaging in patients with suspected, but not yet proven, "acute cardiac syndrome ACS". Patients are included if they presented to the local Emergency Department with chest pain, but the first tests in the Emergency Department are negative or not clearly indicative of cardiac ischemia. For example, the first lab value Troponin T is negative or borderline elevated; or the first ECG is not clearly indicative of ischemia. The standard procedure for these patients is to wait 4-6 hours and then repeat the test; if they continue to be negative, the patients are discharged home, if the have become positive, an invasive coronary artery angiography has to be performed. We think, that a CMR study can shorten the time needed to make the decision of either "discharge" or "admit to CCU and perform a coronary artery angiography". CMR has been shown to be the gold standard for heart function (thus, can see even subtle wall motion abnormalities), for tissue characterization (so-called T2-weighted images can identify tissue edema (swelling); perfusion images can identify areas with reduced blood supply; late enhancement images can safely identify fibrotic or irreversibly damaged tissue) and can even be used to stress the patients to exclude a critical or non-critical narrowing of coronary arteries.

The primary endpoint of this study will be the impact of CMR on the time-to-decision in these patients.

It should be possible to a) identify all patients WITH an acute infarct by CMR and send them to a cath lab sooner compared to waiting for a second test; b) identify all patients WITHOUT an acute infarct and c) perform a stress test in those patients to exclude severe coronary artery disease.

DETAILED DESCRIPTION:
Background

Unstable angina (UA) and non-ST-elevation myocardial infarction (NSTEMI) are serious forms of acute coronary syndromes1. They require rapid clinical assessment, diagnosis and therapeutical intervention. A delay in the diagnosis and a delay in treatment may lead to serious complications such as ventricular arrhythmias, heart failure and sudden cardiac death. In NSTEMI, time delay to diagnosis might lead to irreversible loss of salvageable myocardium.

The current recommendations of the American Heart Association for the management of patients with UA/ NSTEMI rely on the patient's symptoms, ECG changes and serum markers (Troponin) 1. The algorithm for diagnosis and therapy is straight-forward for patients presenting with positive Troponin and/ or ongoing ECG changes; however, an up to 8 hours delay occurs in a patient presenting with chest pain, but without diagnostic ECG changes and negative Troponins (figure 1). During this period, repeat ECGs are recommended to observe changes, and the Troponin test will be repeated at 8 hours.

This delay in diagnosis and treatment might be abbreviated by the diagnosis of UA/NSTEMI with the help of cardiac MRI.

A growing body of evidence supports the capability of MRI to diagnose and rule out UA/ NSTEMI:

In 2003, Kwong et al could show that CMR has not only a high sensitivity and specificity for detecting acute coronary syndromes in the Emergency Room, but it also was the strongest predictor of acute coronary syndromes as compared to ECG, Troponin and a TIMI risk score ≥3. The method appeared suitable for triage of patients presenting with chest pain to the Emergency Room; it was also found to be very safe2. In another study, Plein et al found that CMR could be useful to diagnose coronary artery disease with high sensitivity and specificity in patients presenting to the Emergency Room with chest pain3. Furthermore, it was recently shown that in patients presenting to the ER with chest pain, in whom negative Troponin tests had excluded an acute coronary syndrome, an adenosine stress CMR study was a very powerful predictor of adverse outcomes if positive for perfusion deficits, and a powerful negative predictor if no perfusion deficits were found4.

CMR can visualize irreversible myocardial injury, even if those lesions affect as little as less than 2 grams of myocardial tissue5. Our own data show that CMR is an accurate tool to diagnose acute myocardial infarcts, when T2-weighted imaging for the detection of acute edema is used in conjunction with imaging for irreversible injury6; we also showed that irreversible myocardial injury can be detected as soon as 1 hour after infarction7.

Although it has been shown that CMR can diagnose UA/ NSTEMI2, 3 as well as rule those out with an excellent negative predictive and prognostic value4, it has not been shown whether CMR can lead to a shortening of time-to-diagnosis. It has also not been studied yet, whether or not the incorporation of CMR into the diagnostic pathway would be cost-efficient.

Hypothesis:

Cardiac MRI can shorten the time to diagnosis of acute coronary syndromes in patients presenting with a differential diagnosis of UA/NSTEMI, in whom the initial ECG and Troponin tests are non-diagnostic.

The implementation of CMR into the diagnostic pathway is cost efficient.

Methods:

We will examine patients admitted to the ER with chest pain suggestive of a first acute coronary syndrome. If the initial ECG and Troponin tests are inconclusive and the patient is supposed to wait for a second Troponin test, an urgent CMR study will be performed to diagnose UA/NSTEMI (see figure 2).

The time will be measured from the initial Troponin test to the second decisive Troponin test (control variable). The time will as well be measured from the first Troponin test to the result of the CMR test (test variable).

In patients with a negative CMR study, the CMR study will be extended by a stress perfusion study, and the time will be measured from first negative Troponin to the result of the stress test (test variable). In patients in whom the second Troponin returns negative, and a conventional stress test is scheduled for further diagnostic work-up (independent of the CMR test), the time from the first Troponin to the result of the stress test will be measured.

The CMR study will be performed to assess

1. LV function (global and regional function)
2. Myocardial edema
3. Myocardial perfusion at rest
4. Myocardial infarction
5. If all of the above do not show any pathological result: adenosine stress perfusion

The following protocol will be used for the CMR study:

* Localizer
* LV function in multiple long axes
* T2w STIR in 3 short axis views
* BOLD study in 3 short-axis views
* Rest perfusion study in 3 long axes and 1 short axis view
* Late enhancement study
* If all of the above do not show any pathological result: stress perfusion study with adenosine in 3 long axes and 1 short axis views

The study will be rated positive for an Acute Coronary Syndrome if any one or more of the following will be present:

* Regional wall motion abnormality (in the presence of late enhancement: regional wall motion abnormality in conjunction with positive STIR, or regional wall motion abnormality exceeding the area of late enhancement)
* Regional myocardial edema on the STIR images
* Regional perfusion deficit (in presence of late enhancement: regional perfusion deficit exceeding the area of late enhancement)
* If performed: stress-induced perfusion deficit

The CMR study will be positive for coronary artery disease, but without Acute Coronary Syndrome, when the following criteria will be met:

- Late enhancement without corresponding high signal on STIR, and with or without a regional wall motion abnormality corresponding to but not exceeding the area of late enhancement

Inclusion criteria for this study:

1. 18+ years of age, informed consent obtained
2. Chest pain, suggestive of coronary artery disease, plus at least one more point from the TIMI risk score (TIMI score ≥2)
3. Troponin is negative on 1st draw; based on the Emergency Room Physician's discretion, a 2nd Troponin draw is indicated and pending

Exclusion criteria:

1. ST elevation on ECG, new Q-waves or dynamic ST-segment changes, 2nd or 3rd degree AV-block
2. Unstable patients
3. PCI or myocardial infarction within 3 months
4. Ferromagnetic objects precluding MRI imaging (e.g., pacemaker, defibrillator, cerebral aneurysm clip, metal in eye, insulin pumps, neural stimulators, cochlea implants)
5. Pregnancy
6. Extreme claustrophobia
7. Asthma
8. Inability to lie flat

Endpoints:

Primary Endpoint:

The difference between

1. the Time to diagnosis, measured from the first negative Troponin to the publication of the CMR study report and
2. the Time to diagnosis, measured from the first negative Troponin to the publication of the result of the second Troponin test

Secondary Endpoints:

1. The difference in time to decision for invasive coronary angiography, based on

   1. time to decision based on the CMR test versus
   2. time to decision if the CMR result is neglected and the decision is taken based on the second Troponin test
2. In patients with a negative diagnosis of UA/ NSTEMI, the difference in the time to decision to discharge the patient from the hospital, based on

   1. time to decision based on a negative CMR test
   2. time to decision if the CMR test is neglected and the decision is taken based on a second negative Troponin ± a second negative stress test
3. For 1 and 2, a cost analysis will be performed, assessing total hospital costs for diagnostic algorithms including and excluding CMR, and taking into consideration the costs for CMR, other diagnostic tests and duration of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

1. 18+ years of age, informed consent obtained
2. Chest pain, suggestive of coronary artery disease, plus at least one more point from the TIMI risk score (TIMI score ≥2)
3. Troponin is negative on 1st draw; based on the Emergency Room Physician's discretion, a 2nd Troponin draw is indicated and pending

Exclusion Criteria:

1. ST elevation on ECG, new Q-waves or dynamic ST-segment changes, 2nd or 3rd degree AV-block
2. Unstable patients
3. PCI or myocardial infarction within 3 months
4. Ferromagnetic objects precluding MRI imaging (e.g., pacemaker, defibrillator, cerebral aneurysm clip, metal in eye, insulin pumps, neural stimulators, cochlea implants)
5. Pregnancy
6. Extreme claustrophobia
7. Asthma
8. Inability to lie flat

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The difference between the Time to diagnosis, measured from the first negative Troponin to the publication of the CMR study report | prospective

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Strohm, MD, FESC, Principal Investigator — University of Calgary
Locations (1):
- Stephenson CMR Centre at Foothills Medical Centre, University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Background] Braunwald E, Antman EM, Beasley JW, Califf RM, Cheitlin MD, Hochman JS, Jones RH, Kereiakes D, Kupersmith J, Levin TN, Pepine CJ, Schaeffer JW, Smith EE 3rd, Steward DE, Theroux P, Gibbons RJ, Alpert JS, Faxon DP, Fuster V, Gregoratos G, Hiratzka LF, Jacobs AK, Smith SC Jr; American College of Cardiology; American Heart Association. Committee on the Management of Patients With Unstable Angina. ACC/AHA 2002 guideline update for the management of patients with unstable angina and non-ST-segment elevation myocardial infarction--summary article: a report of the American College of Cardiology/American Heart Association task force on practice guidelines (Committee on the Management of Patients With Unstable Angina). J Am Coll Cardiol. 2002 Oct 2;40(7):1366-74. doi: 10.1016/s0735-1097(02)02336-7. No abstract available. PMID 12383588
- [Background] Kwong RY, Schussheim AE, Rekhraj S, Aletras AH, Geller N, Davis J, Christian TF, Balaban RS, Arai AE. Detecting acute coronary syndrome in the emergency department with cardiac magnetic resonance imaging. Circulation. 2003 Feb 4;107(4):531-7. doi: 10.1161/01.cir.0000047527.11221.29. PMID 12566362
- [Background] Plein S, Greenwood JP, Ridgway JP, Cranny G, Ball SG, Sivananthan MU. Assessment of non-ST-segment elevation acute coronary syndromes with cardiac magnetic resonance imaging. J Am Coll Cardiol. 2004 Dec 7;44(11):2173-81. doi: 10.1016/j.jacc.2004.08.056. PMID 15582315
- [Background] Ingkanisorn WP, Kwong RY, Bohme NS, Geller NL, Rhoads KL, Dyke CK, Paterson DI, Syed MA, Aletras AH, Arai AE. Prognosis of negative adenosine stress magnetic resonance in patients presenting to an emergency department with chest pain. J Am Coll Cardiol. 2006 Apr 4;47(7):1427-32. doi: 10.1016/j.jacc.2005.11.059. Epub 2006 Mar 20. PMID 16580532
- [Background] Schulz-Menger J, Gross M, Messroghli D, Uhlich F, Dietz R, Friedrich MG. Cardiovascular magnetic resonance of acute myocardial infarction at a very early stage. J Am Coll Cardiol. 2003 Aug 6;42(3):513-8. doi: 10.1016/s0735-1097(03)00717-4. PMID 12906982
- [Background] Ricciardi MJ, Wu E, Davidson CJ, Choi KM, Klocke FJ, Bonow RO, Judd RM, Kim RJ. Visualization of discrete microinfarction after percutaneous coronary intervention associated with mild creatine kinase-MB elevation. Circulation. 2001 Jun 12;103(23):2780-3. doi: 10.1161/hc2301.092121. PMID 11401931
- [Background] Abdel-Aty H, Zagrosek A, Schulz-Menger J, Taylor AJ, Messroghli D, Kumar A, Gross M, Dietz R, Friedrich MG. Delayed enhancement and T2-weighted cardiovascular magnetic resonance imaging differentiate acute from chronic myocardial infarction. Circulation. 2004 May 25;109(20):2411-6. doi: 10.1161/01.CIR.0000127428.10985.C6. Epub 2004 May 3. PMID 15123531
- See also: Libin Institute of Alberta — http://www.libin.ucalgary.ca/